CLINICAL TRIAL: NCT05348447
Title: Randomized Trial of Intercostal Nerve Cryotherapy in Patients Undergoing Minimally Invasive Pulmonary Resection
Brief Title: Intercostal Nerve Cryotherapy in Patients Undergoing Minimally Invasive Pulmonary Resection
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other)
Collaborators: AtriCure, Inc. (Industry)
Responsible Party: Principal Investigator, Benny Weksler, MD, System Chief of Thoracic Surgery, Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-238
Record Dates: First submitted 2022-04-15; First posted 2022-04-27 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Cryotherapy Effect; Pain, Postoperative
Keywords: pulmonary; resection; cryotherapy
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Masking Description: participants will be blinded to treatment group and will be sedated (part of standard of care surgery) at the time the treatment occurs
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Cryoanalgesia with standard of care pain control (Experimental): subjects will receive standard of care pain control + cryoanalgesia in the intercostal spaces during routine surgery
  Interventions: Device: cryoanalgesia; Other: Standard of Care Pain Control
- Standard of care pain control (Active Comparator): subjects will receive standard of care pain control only
  Interventions: Other: Standard of Care Pain Control

INTERVENTIONS:
Device: cryoanalgesia — intraoperative intercostal nerve freezing for post-operative pain control
  Arms: Cryoanalgesia with standard of care pain control
Other: Standard of Care Pain Control — Standard of Care Pain Control Post-operatively

SUMMARY:
This is a research study designed to test whether a treatment called Intercostal Nerve Cryotherapy is an effective way to help control post-surgical pain for patients undergoing minimally invasive pulmonary resection.

There are two treatment groups in this study, a cryotherapy group and control group. Cryotherapy is a method of controlling pain by freezing nerves between the ribs that would transmit pain impulses to the brain.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 year and older.
2. Undergoing elective minimally invasive (VATS or robotic) lung resection for nodules (wedge resection, segmentectomy, lobectomy).
3. Performance status of 1 or 2.

Exclusion Criteria:

1. Patients with ejection fraction less than 40%
2. Patients with creatinine greater than 1.5.
3. Patients with Child's B or C cirrhosis
4. Patients on chronic narcotics for other reasons
5. Patients diagnosed with fibromyalgia
6. Patients who had previous thoracic surgery on the same side.
7. Patients who cannot communicate in English.
8. Patients unable to provide informed consent for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-07-07 (Estimated)

PRIMARY OUTCOMES:
Total morphine dose | to discharge (up to 14 days)
  total milligrams (mg) of morphine received during hospitalization
Pain control | to discharge (up to 14 days)
  Pain level, as assessed by visual analog scale (rating 0-10), with 0 being no pain to 10 being worst pain, with higher scores meaning a worse outcome

SECONDARY OUTCOMES:
pulmonary complications | through 1 year
  Pulmonary complications as defined by the Society of Thoracic Surgeons database
pain control | 2 weeks and 3 months post-operatively
  Pain level, as assessed by visual analog scale (rating 0-10), with 0 being no pain to 10 being worst pain, with higher scores meaning a worse outcome
total morphine equivalent dose of narcotics | 2 weeks and 3 months post-operatively
  total dose (e.g. milligrams) assessed by the number of pills taken by patients postoperatively
Presence of neuropathy in the surgical site | 2 weeks, 3 months, 6 months and 1 year postoperatively
  physician will assess by modified treatment-induced neuropathy scale (0-10), with higher scores meaning a worse outcome; The modified questionnaire will assess the following symptoms and ask patients to score those symptoms from 0 (not present) to 10 (unbearable):
  * Numbness at or near the incision site (including chest wall)
  * Tingling at or near the incision site
  * Pain at or near the incision site
  * Hot or burning sensation at or near the incision site
  * Feeling of coldness at or near the incision site
Incentive Spirometer Volume | to discharge (up to 14 days)
  The highest number (breath volume) achieved on exhalation using the incentive spirometer
Hospital length of stay | to discharge (up to 14 days)
  Number of days spent in hospital postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- AHN Allegheny General Hospital, Pittsburgh, Pennsylvania, United States